CLINICAL TRIAL: NCT07233681
Title: Comparison of Serratus Posterior Superior Intercostal Plane Block With Combination of Suprascapular and Infraclavicular Nerve Blocks in Postoperative Analgesia Management in Arthroscopic Shoulder Surgery
Brief Title: Comparison of SPSIPB With SSB and ICB Combination in Arthroscopic Shoulder Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Oguz Gundogdu, Associate Professor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2024-01/07
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Pain After Shoulder Surgery; Shoulder Arthroscopic Surgery
Keywords: suprascapular nerve block; infraclavicular nerve block; Serratus posterior superior intercostal plane block; postoperative pain; arthroscopic shoulder surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of SSB and ICB (Active Comparator): Immediately after anesthesia induction, anterior suprascapular nerve block (SSB) and infraclavicular brachial plexus block (ICB) will be performed on the ipsilateral side with the patient supine. For ICB, a high-frequency linear ultrasound probe is placed sagittally over the lateral infraclavicular fossa, medial to the coracoid process and caudal to the clavicle. The needle is inserted below the clavicle, directed cephalad-to-caudal through the pectoralis major and minor toward the posterior aspect of the axillary artery, and 15 mL of 0.25% bupivacaine is injected. For SSB, the probe is positioned over the supraclavicular fossa in a sagittal oblique plane to visualize the subclavian artery and brachial plexus. The suprascapular nerve is identified beneath the omohyoid muscle, the needle is advanced in-plane from lateral to medial, and 10 mL of 0.25% bupivacaine is administered.
  Interventions: Procedure: suprascapular nerve block
- SPSIPB (Active Comparator): The ultrasound probe was placed 2-3 cm medial to the scapular spine to visualize the trapezius, rhomboid major, and serratus posterior superior muscles. At the level of the 2nd-3rd ribs, a needle was advanced into the plane between the serratus posterior superior muscle and the ribs. After confirming negative aspiration, 30 mL of 0.25% bupivacaine was injected. The block was performed unilaterally, targeting the shoulder undergoing surgery.
  Interventions: Procedure: Serratus posterior superior intercostal plane block

INTERVENTIONS:
Procedure: suprascapular nerve block — Suprascapular nerve block (SSB): 10ml of 0.25% bupivacaine was injected around the suprascapular nerve beneath the omohyoid muscle.
  Infraclavikular nerve block(ICB): The needle is inserted below the clavicle, directed cephalad-to-caudal through the pectoralis major and minor toward the posterior aspect of the axillary artery, and 15 mL of 0.25% bupivacaine is injected
  Arms: Combination of SSB and ICB
Procedure: Serratus posterior superior intercostal plane block — Serratus posterior superior intercostal plane block (SPSIPB): 30 ml of 0.25% bupivacaine was injected into the plane between the serratus posterior superior muscle and the ribs.
  Arms: SPSIPB

SUMMARY:
The aim to compare postoperative analgesic requirements between patients undergoing arthroscopic shoulder surgery who received either the SSB-ICB combination or SPSIPB, and to determine whether one technique has superiority over the other.

DETAILED DESCRIPTION:
Patients were divided into two randomized groups: Group 1 (SSB+ICB combination group, n=15) and Group 2 (SPSIPB group, n=15). All patients will receive the same standard general anesthesia per hospital protocol. All blocks will be applied with the same ultrasonography and block equipment, and by the same physician. Before the anesthesia induction, ipsilateral diaphragmatic excursion will be measured via Ultrasonography (USG). After the anesthesia induction, patients in Group 1 will receive anterior suprascapular nerve block (SSB) with 10 mL of 0.25% bupivacaine and infraclavicular brachial plexus block (ICB) with 15 mL of 0.25% bupivacaine (with a total volume of 25 mL). Patients in Group 2 will receive serratus posterior superior intercostal plane block (SPSIPB) with 30 mL of 0.25% bupivacaine. All patients will receive Paracetamol 1gr and Dexketoprofen 50mg intravenous (IV) 10 minutes prior to skin closure. After 30 minutes of emergence from anesthesia (upon reaching 9 points on modified Aldrete scoring), ipsilateral diaphragmatic excursion will be assessed again. Pre- and postblock excursion differences will be recorded. Routine analgesic procedure consisting of 3x1gr Paracetamol and 2x50mg Dexketoprofen will be followed postoperatively for 24 hours. Numeric Rating Scale (NRS) will be used to assess postoperative pain on 1st, 6th, 12th, 18th and 24th hours after the surgery. Quality of Recovery-15 Patient Survey will be done both preoperatively for a baseline score, and postoperatively at 24th hour to assess the quality of recovery from the patients' view. Tramadol 50mg IV will be administered as a rescue analgesic for all patients if NRS score is higher than 4. Total Tramadol consumption will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients older than 18 years of age who underwent arthroscopic shoulder surgery under general anesthesia and were American Society of Anesthesiologists (ASA) I-II-III according to the ASA risk classification.

Exclusion Criteria:

* patients who did not give consent,
* patients with coagulopathy,
* patients with signs of infection at the block application site,
* patients using anticoagulants,
* patients with local anesthetic drug allergies,
* patients with unstable hemodynamics,
* patients who could not cooperate during postoperative pain assessment
* patients diagnosed with frozen shoulder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | 24 hours after surgery
  Numeric Rating Scale (NRS): The patient selects a number between 0, representing "no pain," and 10 or 100, representing "unbearable pain." This method is highly sensitive and is one of the most commonly used pain scoring tools.
Total tramadol consumption | 24 hours after surgery
  Total postoperative analgesic (tramadol) requirement was recorded in the unit as "milligrams".

SECONDARY OUTCOMES:
Diaphragm Excursion Difference | Preoperatively, immediately before anesthesia induction, and postoperatively, 30 minutes after emergence from anesthesia (when a modified Aldrete score of 9 is reached)
  Ipsilateral diaphragmatic movement will be assessed both immediately before anesthesia induction in the preoperative period and 30 minutes after emergence from anesthesia (when a modified Aldrete score of 9 is reached). A change of up to 25% in diaphragmatic movement indicates no nerve involvement, a change between 25% and 75% indicates partial involvement, and a change exceeding 75% indicates complete phrenic nerve blockade.
Quality of Recovery-15 Patient Questionnaire (QoR-15) | 24th hour after surgery
  The widespread use of minimally invasive procedures to reduce postoperative morbidity and mortality, combined with the implementation of Enhanced Recovery After Surgery (ERAS) protocols, has increased overall interest in the postoperative recovery period and the assessment of outcomes. To address emerging needs in this field, new tools prioritizing patient satisfaction have been developed alongside traditional scales that measure classic parameters. Among these, the Quality of Recovery-15 (QoR-15) patient questionnaire stands out as one of the most up-to-date and reliable instruments. The questionnaire is administered both preoperatively, to record the patient's baseline, and 24 hours after surgery. Higher scores indicate better postoperative recovery quality, with possible scores ranging from 0 to 150.

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Cumhuriyet University, Sivas, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Auyong DB, Hanson NA, Joseph RS, Schmidt BE, Slee AE, Yuan SC. Comparison of Anterior Suprascapular, Supraclavicular, and Interscalene Nerve Block Approaches for Major Outpatient Arthroscopic Shoulder Surgery: A Randomized, Double-blind, Noninferiority Trial. Anesthesiology. 2018 Jul;129(1):47-57. doi: 10.1097/ALN.0000000000002208. PMID 29634491
- [Result] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Sakul BU, Korkmaz AO, Bozkurt NN, De Cassai A, Torres AJ, Elsharkawy H, Alici HA. Serratus Posterior Superior Intercostal Plane Block: A Technical Report on the Description of a Novel Periparavertebral Block for Thoracic Pain. Cureus. 2023 Feb 3;15(2):e34582. doi: 10.7759/cureus.34582. eCollection 2023 Feb. PMID 36883093